CLINICAL TRIAL: NCT00655291
Title: Multicenter, Randomized, Double-Blind, Parallel Group, Placebo-Controlled Study of the Analgesic Efficacy of XP20B in Subjects With Pain Following Bunionectomy Surgery
Brief Title: Efficacy of XP20B Following Bunionectomy Surgery
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Xanodyne Pharmaceuticals (Industry)
Responsible Party: Caroline Masoner/Clinical Trial Manager, Xanodyne Pharmaceuticals
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: XP20B-301
Record Dates: First submitted 2008-04-03; First posted 2008-04-09 (Estimated); Last update posted 2008-10-08 (Estimated); Status verified 2008-10

CONDITIONS: Acute Pain
Keywords: pain
MeSH Terms: conditions — Acute Pain; Pain

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Placebo Comparator)
  Interventions: Drug: Placebo
- B (Experimental)
  Interventions: Drug: XP20B

INTERVENTIONS:
Drug: XP20B
  Arms: B
Drug: Placebo
  Arms: A

SUMMARY:
The purpose of this study is to determine if XP20B is an effective treatment for the relief of pain following bunionectomy surgery.

ELIGIBILITY:
Inclusion Criteria:

* having undergone bunionectomy surgery
* having achieved the requisite level of pain

Exclusion Criteria:

* pregnant or lactating
* history of substance abuse
* clinically significant condition or lab abnormality
* taken any prohibited medications
* gastrointestinal bleeding or history of

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 190 (Estimated)
Dates: Start 2008-04; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
Average pain over a fixed dosing period | Multiple-day

SECONDARY OUTCOMES:
multiple pain assessments over a fixed dosing period | Multiple-day
Rescue medication use | Multiple-day
Safety evaluations | Multiple-day

CONTACTS AND LOCATIONS:
Overall Officials: Keith Moore, PharmD — Xanodyne Pharmaceuticals
Locations (6):
- United States (6):
  - Investigatve Site, Anaheim, California
  - Investigative Site, Owings Mills, Maryland
  - Investigative Site, Austin, Texas
  - Investigative Site, Houston, Texas
  - Investigative Site, San Marcos, Texas
  - Investigative Site, Salt Lake City, Utah